CLINICAL TRIAL: NCT00613769
Title: A Prospective, Randomized, Blind, Multicenter Trial Comparing Orally Administered Trimethoprim-sulfamethoxazole With Intravenously Administered Cefuroxime and Metronidazole as Prophylaxis of Infection Following Elective Colorectal Surgery
Brief Title: Orally Administered Trimethoprim-sulfamethoxazole and Metronidazole as Prophylaxis of Infection Following Elective Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Halmstad County Hospital (Other)
Responsible Party: Principal Investigator, Claes Hjalmarsson, MDPhD, Halmstad County Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TSM; EudraCT number 2006-006575-20
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Infection Prophylaxis in Colo Rectal Surgery
Keywords: Surgical site infections
MeSH Terms: conditions — Surgical Wound Infection | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Metronidazole; Cefuroxime

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ordinary per operative prophylaxis (Active Comparator): cefuroxime(1500mg) i.v.+ metronidazole (1500mg)i.v.given at the time point of induction of anesthesia
  Interventions: Drug: cefuroxime and metronidazole
- Per oral alternative (Experimental): Trimethoprim-sulfamethoxazole(160mg/800mg)p.o.+metronidazole (1200mg)p.o.given 06.00 am on the day of operation
  Interventions: Drug: trimethoprim-sulfamethoxazole + metronidazole

INTERVENTIONS:
Drug: trimethoprim-sulfamethoxazole + metronidazole — trimethoprim-sulfamethoxazole (160mg/800mg)p.o.+ metronidazole (1200mg)p.o.
  Arms: Per oral alternative
Drug: cefuroxime and metronidazole — cefuromime 1500mg i.v. + metronidazole 1500mg i.v.
  Arms: ordinary per operative prophylaxis

SUMMARY:
The current standard Swedish infection prophylaxis in colorectal surgery is intravenously administered cefuroxime and metronidazole. this combination is well studied. The disadvantages of the regimen is "collateral damage" resulting from treatment with a cephalosporine and that the combination also serves as the first line of treatment for abdominal surgical infections.

Serval Swedish surgical departments have for some years used a combination of orally administered trimethoprim-sulfamethoxazole and metronidazole.

The combination is economical and believed to be effective but hitherto the outcome have not been properly researched.

The aim of this study is to compare the efficacy of these two regimens in the prevention of infection after elective colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Planned clean/clean-contaminated colorectal resection will be performed
* Understand spoken and written swedish language

Exclusion Criteria:

* Hypersensibility to the test or control drug
* Severe liver failure
* Blood dyscrasia
* Ileus or gastric retention
* Current visceral perforation
* Current treatment with antibiotics
* Current treatment with steroids
* Cytotoxic or radiation therapy within 4 weeks of the planned operation
* Active IBD (inflammatory bowel disease)
* Incapability to swallow tablets
* Other study interfering with this study
* Current pregnancy
* Bad regulated diabetes
* Current enterocutaneous or colocutaneous fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1073 (Actual)
Dates: Start 2007-09; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Cutaneous-,subcutaneous and intraabdominal infections | 4 weeks

SECONDARY OUTCOMES:
Non infectious wound complications | 4 weeks
Complications to the anastomosis | 4 weeks
Adverse reaction of given drug | 4 weeks
Other post operative infections | During hospital stay
Septicaemia | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claes Hjalmarsson, MD,PhD, Principal Investigator — Department of Surgery and Oncology, Halland Hospital Halmstad, 301 85 Halmstad, Sweden
Locations (6):
- Sweden (6):
  - Department of Surgery, University hospital Sahlgrenska/Östra, Gothenburg
  - Department of Surgery and oncology, Halland Hospital in Halmstad, Halmstad
  - Department of surgery, Community Hospital i Karlskrona, Karlskrona
  - Vrinnevi hospital, Norrköping
  - Department of surgery, Skövde
  - Department of Surgery, NU-hospitals, Uddevalla